CLINICAL TRIAL: NCT01495663
Title: A Phase 1, Multi-Center, Open-Label, Dose Escalation Study of I-131-CLR1404 in Subjects With Relapsed or Refractory Advanced Solid Malignancies
Brief Title: Dose Escalation Study of I-131-CLR1404 in Subjects With Cancer That Does Not Respond to Treatment or Has Returned
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCL-10-001
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Cancer
Keywords: refractory; relapsed; non-small cell lung cancer; triple-negative breast cancer; soft tissue sarcoma; colorectal cancer; esophageal cancer; prostate cancer; ovarian cancer
MeSH Terms: conditions — Neoplasms; Recurrence; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Sarcoma; Colorectal Neoplasms; Esophageal Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms | interventions — CLR1404

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group (Other): I-131-CLR1404
  Interventions: Drug: I-131-CLR1404

INTERVENTIONS:
Drug: I-131-CLR1404 — Description:
  * Dosimetry: IV, 5 mCi, single dose, 6-day duration
  * Therapy: IV, starting dose level of 12.5 mCi/m2, single dose, 56-day duration with follow up to one year
  Other Names: 18-(p-[I-131]-iodophenyl)octadecyl phosphocholine

SUMMARY:
The purpose of this study is to determine the recommended dose of I-131-CLR1404, a radiolabeled therapy compound, for treating subjects with cancer that does not respond to treatment or has returned. The identified recommended dose in this study will be used as the optimal dose of I-131-CLR1404 in subsequent clinical trials conducted for later phase clinical development.

Subjects who meet study entry criteria will receive I-131-CLR1404. For each subject, the study will be conducted in two phases, dosimetric and therapy. In the dosimetric phase, subjects will receive one 5 mCi dose of the study drug and undergo whole body imaging on on the day of infusion and on post-infusion days 1, 2, 3, and 6 for assessment of biodistribution of I-131-CLR1404. If normal and expected biodistribution are demonstrated, the subject will begin the therapy phase. In the therapy phase, the first cohort of subjects will receive a dose of 12.5 mCi/m2. Dose escalation in subsequent cohorts will initially be in increments of 12.5 mCi/m2. Subjects will be followed and observed for unacceptable toxicity through 56 days after the therapy dose infusion with follow-up for up to one year.

All subjects will be prescribed thyroid protection medication to be taken 24 hours prior to injection of the dosimetric dose, and continuing for 14 days after the administration of the therapy dose.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory advanced solid malignancy or choice not to pursue standard treatment. Tumor types allowed: non-small cell lung, triple negative breast, soft tissue sarcoma, colorectal, gastric, esophageal, prostate, ovarian cancer
* ≥ 1 lesion that qualifies as a "target lesion" based on RECIST 1.1
* Ambulatory w/ECOG performance status 0 to 2 and estimated life expectancy ≥ 4 mo.
* 18 years or older
* Judged by Investigator to have initiative and means to be compliant with protocol and w/n geographical proximity to make required study visits
* Ability to read, understand and provide written informed consent for initiation of any study related procedures (subject or legal representative)
* Brain metastasis acceptable if clinical condition stable ≥ 1 mo. Subjects with brain metastasis requiring steroids must have been on a stable or tapering dose of corticosteroids ≥ 1 mo. prior to enrollment
* Negative serum pregnancy test w/n 24 hours of enrollment (Female subjects of childbearing potential)
* Agreement to use effective contraception method (oral contraceptives, double-barrier methods, intrauterine device, Norplant, Depo-Provera) during study and 90 days following last dose

Exclusion Criteria:

* Subject or physician plans concomitant chemotherapy, therapeutic radiation and/or biological treatment for cancer including immunotherapy while on study. Localized palliative radiation therapy for bone pain allowed if clinically indicated. Ongoing hormonal therapy may be continued
* Received > 3 previous cytotoxic chemotherapy regimens
* Received > 25% of total bone marrow irradiated, total body or hemi-body irradiation or prior radioisotope therapy (except for benign thyroid disease)
* Diffuse lung disease or interstitial spread of carcinoma
* Prior radiation therapy or chemotherapy w/n 4 weeks of study start
* Extradural tumor in contact with spinal cord or tumor located where swelling in response to therapy may impinge upon spinal cord
* Other active medical condition or organ disease that may compromise safety or interfere with safety and/or outcome evaluation of study drug
* Laboratory abnormalities, including but not limited to: WBC < 3000/uL, Absolute neutrophil count < 1500/uL, Platelets < 150,000/uL, Hemoglobin ≤ 9.0 gm/dL, Total bilirubin > 1.5 x upper limit of normal for age, SGOT or SGPT > 3 x upper limit of normal for age if no liver metastases or > 5 x upper limit of normal for age in the presence of liver metastases, Serum creatinine > 1.5 x upper limit of normal for age, INR ≥ 2.0, 2+ proteinuria or casts indicative of intrinsic renal disease
* Treatment with investigational drug, investigational biologic, or investigational therapeutic device w/n 28 days of initiating study treatment
* Received severely marrow toxic drugs (eg nitrosoureas, mitomycin)
* Received blood transfusions or hematopoietic growth factor therapy w/n 30 days of study start
* Received prior stem cell transplantation
* Clinically significant cardiac co-morbidities including congestive heart failure (New York Heart Association class III-IV heart disease), left ventricular ejection fraction < 40%, unstable angina pectoris, serious cardiac arrhythmia requiring medication or pacemaker, myocardial infarction within past 6 months
* Concurrent or recent (w/n 1 month) use of thrombolytic agents or full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters). Therapy with low-molecular weight heparin is acceptable as long as INR < 2.0
* Uncontrolled hypertension as defined by systolic blood pressure > 150 mm/Hg, diastolic blood pressure > 100 mm/Hg or uncontrolled diabetes that would compromise subject safety or interfere with safety and/or outcome evaluation of study drug
* Grade II-IV peripheral vascular disease or peripheral vascular surgery w/n past year
* Major surgery w/n 4 wks. of enrollment
* Poor venous access and unable to receive study drug into a peripheral venous catheter
* Significant traumatic injury w/n past 4 wks.
* Ongoing or active infection requiring antibiotics or with fever >38.1º C (>101º F) w/n 3 days of first scheduled day of dosing
* Receiving concurrent hemodialysis or peritoneal dialysis
* Known positive for HIV, Hepatitis C (active, previously treated or both) or is Hepatitis B core antigen positive
* Pregnant or lactating
* Hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Determination of the recommended dose of I-131-CLR1404 in treating subjects with relapsed or refractory advanced solid malignancies | Until non-tolerated dose is defined; dose escalation descision made upon review of data from a complete cohort (56 days after all subjects in cohort have received therapy infusion)
  Largest administered dose with at most a 20% dose limiting toxicity rate

SECONDARY OUTCOMES:
Expansion of the safety profile of I-131-CLR1404 | Pre-infusion and 6 days after dosimetry infusion; weekly until 56 days after therapy infusion and then monthly for one year
  Assesment by physical examination, vital signs, ECG, laboratory changes over time, and adverse events
Expansion of the pharmacokinetic profile of I-131-CLR1404 | Pre-infusion and 144 hours post-dosimetry infusion; pre-infusion, 5, 15, 60 minutes, 5, 24, 72 hours, 6, 14, 21, 28, 35, 42, 49 and 56 days post-therapy infusion
  Determination of the following pharmacokinetic parameters of I-131-CLR1404:
  * Area under the plasma concentration versus time curve (AUC)
  * Maximum (peak) plasma concentration (Cmax)
  * Time required to reduce the plasma concentration to one half its initial value (t1/2)
  * Volume of distribution (Vd)
  * Clearance of the drug from plasma (Cl)
Preliminary antitumor activity of I-131-CLR1404 | Baseline at screening, 56 days post-therapy infusion, every 2 months in follow-up period up to one year
  CT imaging (response and progression will be evaluated using RECIST 1.1) and tumor marker evaluation in subjects with applicable tumors (performed at screening, 28 and 56 days post-therapy infusion)
Tumor dosimetry of I-131-CLR1404 in a subset of subjects with non-hepatic lesions measuring at least 2 cm in one dimension | 72 hours, 6, 14, and 21 days post-therapy infusion
  SPECT or SPECT/CT

CONTACTS AND LOCATIONS:
Overall Officials: Glen Liu, M.D, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin